CLINICAL TRIAL: NCT01212081
Title: Assessment of Cannabis Craving in Schizophrenia Using Virtual Reality
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910462; 10-DA-N462
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2012-11-26

CONDITIONS: Cannabis Use
Keywords: Virtual Reality; Schizophrenia; Cannabis; Assessment; Craving
MeSH Terms: conditions — Schizophrenia; Marijuana Abuse

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Individuals with schizophrenia or schizoaffective disorders have a high prevalence of cannabis use. Understanding some of the environmental factors that maintain cannabis use, such as socially triggered cravings, is a critical step in improving treatment for cannabis dependence. In recent years, virtual reality has been studied to determine whether it can be used to induce craving by using life-like cue settings. Researchers are interested in using virtual reality systems to study cannabis cravings in individuals with schizophrenia.

Objectives:

- To determine if virtual reality cues will elicit cannabis craving in persons with schizophrenia who have a history of cannabis use.

Eligibility:

- Individuals between 18 and 50 years of age who have been diagnosed with schizophrenia or schizoaffective disorders, are on a stable antipsychotic medication, and who have a lifetime history of at least 50 cannabis uses and average cannabis use of once per month.

Design:

* This study involves an initial screening visit, a study visit, and a followup visit.
* Participants will be screened with a medical history and physical examination, and will complete questionnaires about their history of marijuana and other drug use. Participants will also learn how to use the virtual reality equipment at this visit.
* During the study visit, participants will respond to marijuana cues using the virtual reality system while researchers monitor their heart rate, blood pressure, and sweat levels.
* At the followup visit, participants will complete questionnaires about their mood and any cravings for marijuana.

DETAILED DESCRIPTION:
Objective: The use of cannabis is prevalent in people with schizophrenia, and has been linked both to onset of illness and worsening of symptoms. Craving in persons with schizophrenia who use cannabis has not been widely studied. The occurrence of craving may lead to relapse in substance use disorders. Therefore, craving paradigms in people with schizophrenia need to be optimized in order to test new treatments on craving measures in this population. Thus, the purpose of this study is to determine the feasibility and effects of virtual reality cues on craving intensity for cannabis in patients with schizophrenia

Study population: We will enroll 25 persons with a DSM IV diagnosis of schizophrenia who have a lifetime history of at least 50 lifetime uses of cannabis and cannabis use an average of at least once per month (or, if inpatients, average use of once per month prior to hospitalization) with a goal of 16 completers.

Design: This study uses a comparison-controlled, within-subject design. All subjects will undergo a baseline assessment and acclimation period and then participate in an experimental condition in which four cues will be presented in separate rooms in the VR program. These include two cannabis cues and two neutral cues in four different rooms. A follow up session for craving and symptom assessments will occur one week after the experimental session.

Outcome Measures:

At the end of each of the four cues, the Cannabis Craving Scale (CCVAS), Cannabis Attention scale (CAS), the Marijuana Craving Questionnaire-Short Form (MCQ-SF), and a visual analog cigarette craving item will be administered to measure craving during the virtual reality session. The CCVAS and CAS will be projected into the VR environment and participants will respond via hand controller. The MCQ-SF will also be administered, as well as the Mood form , to assess mood, at baseline as well as at the end of each of the 4 cues. Before and after the experimental session participants will also be rated on the Brief Psychiatric Rating Scale (BPRS), Schedule for the Assessment of Negative Symptoms (SANS), side effects, and the State-Trait Anxiety Inventory (STAI). The Immersion Questionnaire and Imagery Realism Presence Questionnaire (PQ) will be given at the conclusion of the experimental session. Before and after the session, as well as during the experiment participants will be monitored for physiological reactivity (heart rate, blood pressure, and skin conductance response) to cues of cannabis use as well as neutral cues measured.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA FOR SCHIZOPHRENIA PATIENTS:

INCLUSION CRITERIA:

1. 18-55 year old males and females
2. Lifetime history of at least 50 cannabis uses and average cannabis use of once per month (or average use of once per month prior to hospitalization, if inpatient)
3. Current DSM-IV diagnosis of schizophrenia or schizoaffective disorder
4. Stable antipsychotic regimen (4 weeks on antipsychotic regimen and 30 days at current dose)
5. Medically healthy as determined by screening criteria
6. Agrees to wear a head mounted display (HMD) for a period of time generally not exceeding 45 minutes

EXCLUSION CRITERIA:

1. DSM-IV diagnosis of active alcohol or substance abuse (besides cannabis or nicotine) in the past 1 month or dependence within the past 6 months
2. Current use of any medication that would interfere with the protocol in the opinion of MAI (dronabinol, varenicline, bupropion, etc)
3. History of head injury, seizures, stroke, or severe motion sickness
4. Positive urine toxicology screen for agents besides cannabis for substances other than cannabis or those used for therapeutic purposes: Participants who have an initial positive urine toxicology screen for substances other than those used for therapeutic purposes or cannabis will have the opportunity to return within two weeks for a second toxicology screen. If at that time the results are again positive, the participant will be excluded.
5. Positive pregnancy test (if female)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-09-26; Study Completion 2012-11-26

PRIMARY OUTCOMES:
Primary measures include the Cannabis Craving Scale, Cannabis Attention Scale, and Marijuana Craving Questionnaire-Short Form, assessed after each cue. Physiological measures (blood pressure, heart rate, skin conductance) are continuously measur...

SECONDARY OUTCOMES:
Secondary measures include the Mood form, assessed at baseline and after each cue, and measures of the virtual reality experience including the Immersion Questionnaire and Imagery Realism Presence Questionnaire, administered following the sessio...

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Heishman, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland, United States

REFERENCES:
- [Background] Addington J, Addington D. Patterns, predictors and impact of substance use in early psychosis: a longitudinal study. Acta Psychiatr Scand. 2007 Apr;115(4):304-9. doi: 10.1111/j.1600-0447.2006.00900.x. PMID 17355521
- [Background] Andreasen NC. Negative symptoms in schizophrenia. Definition and reliability. Arch Gen Psychiatry. 1982 Jul;39(7):784-8. doi: 10.1001/archpsyc.1982.04290070020005. PMID 7165477
- [Background] Bordnick PS, Graap KM, Copp H, Brooks J, Ferrer M, Logue B. Utilizing virtual reality to standardize nicotine craving research: a pilot study. Addict Behav. 2004 Dec;29(9):1889-94. doi: 10.1016/j.addbeh.2004.06.008. PMID 15530734